CLINICAL TRIAL: NCT02357134
Title: High-Flow Oxygen for Exertional Dyspnea in Cancer Patients
Brief Title: High-Flow Oxygen in Reducing Shortness of Breath Caused by Exercise in Patients With Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2014-0971; NCI-2015-00418 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0971 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-01-29; First posted 2015-02-06 (Estimated); Results first posted 2021-06-01 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-11

CONDITIONS: Dyspnea; Malignant Neoplasm
MeSH Terms: conditions — Dyspnea; Neoplasms | interventions — Oxygen; Respiratory Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm I (high-flow oxygen) (Experimental): Patients receive high-flow oxygen via nasal prongs during a structured stationary bicycle exercise session.
  Interventions: Procedure: Oxygen Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (high-flow air) (Experimental): Patients receive high-flow air via nasal prongs during a structured stationary bicycle exercise session
  Interventions: Procedure: Oxygen Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm III (low-flow oxygen) (Active Comparator): Patients receive low-flow oxygen via a nasal cannula during a structured stationary bicycle exercise session.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Respiratory Therapy
- Arm IV (low-flow air) (Active Comparator): Patients receive low-flow air via a nasal cannula during a structured stationary bicycle exercise session.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Respiratory Therapy

INTERVENTIONS:
Procedure: Oxygen Therapy — Receive high-flow oxygen
  Other Names: supplemental oxygen therapy
  Arms: Arm I (high-flow oxygen)
Procedure: Oxygen Therapy — Receive high-flow air
  Other Names: supplemental oxygen therapy
  Arms: Arm II (high-flow air)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Procedure: Respiratory Therapy — Receive low-flow oxygen
  Arms: Arm III (low-flow oxygen)
Procedure: Respiratory Therapy — Receive low-flow air
  Arms: Arm IV (low-flow air)

SUMMARY:
This randomized phase II trial studies how well high-flow oxygen works in reducing difficulty breathing during exercise (exertional dyspnea) in patients with cancer. Dyspnea is linked to decreased lung function, quality of life, and survival. High-flow oxygen is a device that delivers heated and humidified oxygen through the nose. This may be effective in reducing dyspnea, and may help patients' lungs function better and improve their quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Obtain preliminary estimates of the effect size of oxygen and high flow rate on exertional dyspnea (modified Borg Scale adjusted for work rate and baseline dyspnea).

SECONDARY OBJECTIVES:

I. Determine the completion rate of a randomized controlled trial of exertional dyspnea in cancer patients.

II. Obtain preliminary estimates of the effects of oxygen and flow rate on physiologic function (respiratory rate and oxygen saturation) and exercise capacity (work rate and exercise duration).

OUTLINE: All patients undergo a baseline structured exercise session with air. Patients are then randomized to 1 of 4 treatments for a second session approximately 3 days later.

ARM I: Patients receive high-flow oxygen via nasal prongs during a structured stationary bicycle exercise session.

ARM II: Patients receive high-flow air via nasal prongs during a structured stationary bicycle exercise session.

ARM III: Patients receive low-flow oxygen via a nasal cannula during a structured stationary bicycle exercise session.

ARM IV: Patients receive low-flow air via a nasal cannula during structured stationary bicycle exercise session.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer, with evidence of primary or secondary lung involvement
* Average dyspnea Borg Scale >= 4 of 10 with severe exertion over the past week
* Oxygen saturation > 90% on ambient air at time of assessment
* Able to communicate in English or Spanish
* Karnofsky performance status >= 50%
* Seen at Supportive Care, cardiopulmonary center, thoracic radiation oncology or thoracic medical oncology

Exclusion Criteria:

* Resting dyspnea modified Borg Scale > 7 of 10 at enrollment
* Severe obstructive lung disease (forced expiratory volume in 1 second [FEV1]/forced vital capacity [FVC] < 70% post bronchodilator and forced expiratory volume in 1 second < 30% predicted)
* Delirium (i.e., Memorial Delirium Rating Scale > 13)
* History of unstable angina or myocardial infarction in the last week
* Acute pulmonary embolus or pulmonary infarction in the last week
* Thrombosis of lower extremities in the last week
* Acute myocarditis, pericarditis, or endocarditis in the last week
* Symptomatic aortic stenosis or syncope in the last week
* Suspected dissecting aneurysm
* Severe untreated resting arterial hypertension (> 200 mmHg systolic, > 120 mmHg diastolic) at the time of enrollment
* Uncontrolled arrhythmias causing symptoms or hemodynamic compromise in the last week
* Uncontrolled heart failure in the last week
* Pleural effusion requiring thoracentesis within 1 week of study enrollment or scheduled during the study period
* Airway obstruction requiring stenting within 1 week of study enrollment or scheduled during the study period
* Pneumonia requiring antibiotics at the time of study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2015-03-17 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2023-05-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: David Hui, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Hui D, Mahler DA, Larsson L, Wu J, Thomas S, Harrison CA, Hess K, Lopez-Mattei J, Thompson K, Gomez D, Jeter M, Lin S, Basen-Engquist K, Bruera E. High-Flow Nasal Cannula Therapy for Exertional Dyspnea in Patients with Cancer: A Pilot Randomized Clinical Trial. Oncologist. 2021 Aug;26(8):e1470-e1479. doi: 10.1002/onco.13624. Epub 2020 Dec 14. PMID 33289280
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the Supportive Care, Thoracic Radiation Oncology and Thoracic Medical Oncology clinics at MD Anderson Cancer Center, Houston, USA between 3/2015 and 4/2018 .
Pre-assignment Details: A total of 74 participants were enrolled but 45 patients were randomized for this study. 29 patients were not randomized for various reasons (became ineligible or too symptomatic to participate while waiting=14, scheduling conflict=9, exertional dyspnea too low=4, could not complete baseline test due to desaturation=1, hypertension during exercise=1)
Groups:
- High Flow Oxygen: High Flow Oxygen were delivered between 20 and 70 L/min.
- High Flow Air: High Flow Air were delivered between 20 and 70 L/min.
- Low Flow Oxygen: Low Flow Oxygen were delivered at 2 L/min.
- Low Flow Air: Low Flow Air were delivered at 2 L/min
Period: Overall Study
Arm/Group | High Flow Oxygen | High Flow Air | Low Flow Oxygen | Low Flow Air
Started | 11 | 11 | 12 | 11
Completed | 10 | 11 | 12 | 11
Not Completed | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The data is provided for 44 participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | High Flow Oxygen | High Flow Air | Low Flow Oxygen | Low Flow Air | Total
Number analyzed (Participants) | 10 | 11 | 12 | 11 | 44
Age, Continuous [Mean (Full Range); unit: years] | 59 [48 to 72] | 67 [55 to 75] | 63 [51 to 77] | 62 [47 to 73] | 63 [47 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 3 | 5 | 18
  Male | 5 | 6 | 9 | 6 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 2 | 4
  Not Hispanic or Latino | 10 | 10 | 11 | 9 | 40
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 1 | 1 | 5
  White | 7 | 10 | 11 | 10 | 38
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 12 | 11 | 44
Cancer Type [Count of Participants; unit: Participants]
  Mesothelioma | 0 | 0 | 2 | 3 | 5
  Non Small Cell Lung Cancer | 7 | 9 | 7 | 5 | 28
  Small Cell Lung Cancer | 1 | 1 | 2 | 2 | 6
  Other | 2 | 1 | 1 | 1 | 5
Cancer Stage [Count of Participants; unit: Participants]
  Localized | 1 | 3 | 3 | 0 | 7
  Locally advanced | 3 | 4 | 4 | 6 | 17
  Metastatic | 6 | 4 | 5 | 5 | 20
Comorbidities [Count of Participants; unit: Participants]
  COPD | 5 | 3 | 2 | 1 | 11
  Heart Failure | 1 | 1 | 1 | 0 | 3
  Asthma | 1 | 1 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Modified Borg Scale Dyspnea Intensity at Isotime
Description: Assessed Dyspnea using the Modified Borg Scale Dyspnea Intensity that ranges from 0 ("no shortness of breath") to 10 ("worst possible shortness of breath") at Isotime. Measured the mean difference of Modified Borg Scale Dyspnea Intensity at isotime between the second exercise test (in which all patients received Low Flow Oxygen) and the third exercise tests (in which all patients received the assigned intervention).
Time Frame: End of second exercise test and end of third exercise test, approximately up to 12 minutes
Population: The data is provided for 44 participants who completed the study.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | High Flow Oxygen | High Flow Air | Low Flow Oxygen | Low Flow Air
Number analyzed (Participants) | 10 | 11 | 12 | 11
score on a scale | -1.1 [-2.1 to -0.12] | -0.2 [-0.97 to 0.6] | -1.8 [-2.7 to -0.9] | -0.5 [-1.3 to 0.4]

2. Secondary Outcome: Slope of Modified Borg Scale Dyspnea Unpleasantness Over Time During Constant Work Exercise Per Minute (Third Test)
Description: Dyspnea unpleasantness was measured using the Modified Borg Scale Dyspnea Intensity that ranges from 0 ("no shortness of breath") to 10 ("worst possible shortness of breath"). Dyspnea intensity was measured every minute. The number of minutes varied by patient, per test. It was measured as pairwise difference of slope (taking 'low flow air' arm as a reference). This linear mixed model was constructed based on the following: Dyspnea Unpleasantness at third test = Minutes + Study Arm + Study Arm*Minutes + Total work rate + Slope of Dyspnea Unpleasantness and Minutes at Second test + Minutes at second test.
Time Frame: Third exercise test, approximately up to 12 minutes
Population: The data is provided for 44 participants who completed the study.
Measure: Mean (95% Confidence Interval); unit: Units on a scale per minute
Arm/Group | High Flow Oxygen | High Flow Air | Low Flow Oxygen | Low Flow Air
Number analyzed (Participants) | 10 | 11 | 12 | 11
Units on a scale per minute | 0.55 [0.50 to 0.62] | 0.78 [0.71 to 0.87] | 0.59 [0.52 to 0.67] | 0.69 [0.60 to 0.79]

3. Secondary Outcome: Modified Borg Scale Leg Discomfort
Description: Leg discomfort was measured using the Modified Borg Scale Leg discomfort that ranges from 0 ("no discomfort") to 10 ("worst possible discomfort") during the constant work exercise of third test. Leg discomfort was measured every minute. The number of minutes varied by patient, per test. It was measured as pairwise difference of slope (taking 'low flow air' arm as a reference). This linear mixed model was constructed based on the following: Leg Discomfort at third test = Minutes + Study Arm + Study Arm*Minutes + Total work rate + Slope of Leg Discomfort and Minutes at Second test + Minutes at Second test.
Time Frame: Third exercise test, approximately up to 12 minutes
Measure: Mean (95% Confidence Interval); unit: Units on a scale per minute
Arm/Group | High Flow Oxygen | High Flow Air | Low Flow Oxygen | Low Flow Air
Number analyzed (Participants) | 10 | 11 | 12 | 11
Units on a scale per minute | 0.59 [0.53 to 0.64] | 0.91 [0.82 to 0.99] | 0.65 [0.58 to 0.74] | 0.81 [0.71 to 0.91]

4. Secondary Outcome: Exercise Endurance
Description: The Exercise endurance was measured as a mean duration of constant work in minutes during third test. It was measured as pairwise comparison of mean difference of exercise duration (taking 'low flow air' as a reference). This linear mixed model was constructed based on the following: Time at third test = Study Arm + Minutes at Second test. Detail output from the mixed models
Time Frame: End of third exercise test, approximately up to 12 minutes
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | High Flow Oxygen | High Flow Air | Low Flow Oxygen | Low Flow Air
Number analyzed (Participants) | 10 | 11 | 12 | 11
minutes | 10.50 [7.48 to 13.52] | 8.18 [7.03 to 9.34] | 7.58 [6.0 to 9.17] | 7.36 [6.35 to 8.37]

5. Secondary Outcome: Adverse Events
Description: Adverse effects related to supplemental oxygen use were assessed using a numeric rating scale from 0 (not at all) to 10 (worst possible) before and after the study intervention. The mean change was measured before and after the 3rd test ranging between -10 (improvement) and +10 (deterioration).
Time Frame: Before and after 3rd test during intervention phase, approximately up to 12 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High Flow Oxygen | High Flow Air | Low Flow Oxygen | Low Flow Air
Number analyzed (Participants) | 10 | 11 | 12 | 11
units on a scale
  Dry eyes | 0 (0) | 0 (0) | 0.17 (0.94) | 0 (0)
  Dry Nose | 0 (0) | -0.45 (1.21) | -.033 (0.89) | 0.3 (0.67)
  Eye Irritation | -0.1 (0.32) | 0 (0) | 0.33 (1.15) | 0 (0)
  Moisture in nose | 1 (3.8) | 0.73 (1.56) | 0 (1.13) | 1.5 (2.8)
  Nasal Prongs Uncomfortable | -0.3 (0.67) | 0.18 (0.87) | -0.17 (0.94) | 0.3 (0.67)
  Suffocating | 0.1 (1.2) | -0.09 (0.54) | 0.08 (0.29) | 0.4 (0.7)
  Anxious | 0.4 (1.78) | -0.55 (1.29) | 0.17 (0.72) | 0.5 (1.58)
  Difficulty talking | -0.1 (0.57) | 0.09 (0.3) | 0 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: before and after 3rd test during intervention phase, approximately up to 12 minutes
Description: In this protocol, the Adverse events were not measured as an absolute number. It was measured as a numeric rating score from 0 (not at all) to 10 (worst possible). So there are no Adverse events numbers in the Adverse Events section. As per the protocol, Adverse events were considered as a secondary outcome. Please see 'Adverse Events' under 'Outcome Measure.'
Arm/Group | High Flow Oxygen | High Flow Air | Low Flow Oxygen | Low Flow Air
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-17): https://cdn.clinicaltrials.gov/large-docs/34/NCT02357134/Prot_SAP_000.pdf